CLINICAL TRIAL: NCT04174755
Title: Semaglutide's Efficacy in Achieving Weight Loss for Those With HIV
Acronym: SWIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: University of Copenhagen (Other); Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Mallon, Professor of Microbial Diseases, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWIFT Study
Record Dates: First submitted 2019-11-06; First posted 2019-11-22 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Obesity; HIV-1-infection
Keywords: obesity; HIV; weight loss; GLP-1 analogue; immune activation; viral reservoir; gut microbiome
MeSH Terms: conditions — Obesity; Weight Loss | interventions — semaglutide; Standard of Care; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide 0.25/0.5/1 mg plus standard of care (Experimental)
  Interventions: Drug: Semaglutide Injectable Product; Behavioral: Standard of care
- Standard of care alone (Other)
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Drug: Semaglutide Injectable Product — Semaglutide 0.25 mg subcutaneously once weekly for 4 weeks, then Semaglutide 0.5 mg subcutaneously once weekly for 4 weeks, then Semaglutide 1 mg subcutaneously once weekly for 20 weeks. Total treatment duration 28 weeks.
  Other Names: Ozempic
  Arms: Semaglutide 0.25/0.5/1 mg plus standard of care
Behavioral: Standard of care — Diet and exercise advice for 40 weeks
  Other Names: Diet and exercise

SUMMARY:
The prevalence of obesity is rising worldwide, both in low- and high-income countries, including people with HIV (PWH). Semaglutide's efficacy in achieving weight loss in obese PWH is still unexplored. The aim of this study is to assess the efficacy and safety of semaglutide in achieving greater weight loss compared to diet and excercise alone in obese PWH and to explore the effect of semaglutide on the immune function, markers of immune activation, viral reservoir, markers of glucose and lipid metabolism and gut microbiome.

DETAILED DESCRIPTION:
A randomised, controlled, parallel-group, open-label study comparing treatment with the GLP-1 analogue semaglutide in combination with lifestyle interventions to lifestyle interventions alone in obese PWH.

The study will enroll HIV-1 infected patients ≥ 18 years with BMI ≥30kg/m2 or BMI ≥27kg/m2 and hypertension, dyslipidaemia or type 2 diabetes mellitus.

Primary objective: To assess the efficacy of semaglutide as an adjunct to diet and exercise in achieving greater weight loss in obese PWH as compared to diet and exercise alone.

Secondary objectives:

* To explore the effect of semaglutide on markers of immune function and HIV viral reservoirs in obese PWH.
* To explore the effect of semaglutide on markers of glucose and lipid metabolism in obese PWH.
* To explore the effect of semaglutide on markers of inflammation and gut microbial translocation in obese PWH.
* To assess the safety of semaglutide in obese PWH on stable ART.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Be HIV-1 antibody positive as determined by a positive 4th generation Ag/Ab ELISA assay
* Be stable on ART with a viral load suppressed <40 copies/mL for a minimum of 2 years
* Have a CD4 count ≥200 cells/mm3 for a minimum of 1 year
* Have a BMI ≥30kg/m2 or have a BMI ≥27kg/m2 and hypertension, dyslipidaemia or type 2 diabetes mellitus
* Understand the study procedures, be able to comply with the study procedures, and voluntarily agree to participate by giving written informed consent for the trial

Exclusion Criteria:

* Subjects unable to comply with the study protocol or unable to self-administer subcutaneous semaglutide
* History of obesity induced by other endocrine disorders: hypothyroidism, Cushing's syndrome, primary and secondary hypogonadism, hypothalamic disorders, polycystic ovary syndrome, insulinoma
* History of obesity induced by use of anti-psychotic medications known to be associated with weight gain (i.e. olanzapine, clozapine).
* Treatment with GLP-1 receptor agonists (including liraglutide, semaglutide or exenatide), dipeptidyl peptidase-4 (DPP-4) inhibitors or insulin within the last 3 months (including saxagliptin, linagliptin, sitagliptin)
* History of severe renal impairment, as defined by a baseline creatinine clearance <30ml/min
* Individuals with a diagnosis of HIV-associated lipoatrophy/lipodystrophy, based on physician's assessment
* Individuals with severe hepatic impairment (Child Pugh score >9)
* Subjects with active hepatitis B infection (defined as hepatitis B sAg positive) or hepatitis C (defined as hepatitis C Ab and RNA positive) co-infection
* Any active illness (including AIDS-defining illness) which in the opinion of the investigator precludes participation in the study
* History of cancer (apart from treated Kaposi's Sarcoma) and/or receiving chemotherapy or radiotherapy
* Active illicit intravenous drug use
* Subjects concurrently enrolled in another clinical trial of an investigational medicinal product.
* The investigator may decide that a subject cannot proceed in the study if there is any relevant other abnormal results in the screening assessments
* Subjects with any known or suspected hypersensitivity to semaglutide or any of the excipients of semaglutide
* Subjects on another medicinal product prescribed primarily for weight loss e.g. orlistat (see prohibited/cautioned concomitant medications/therapies section)
* For female subjects: pregnancy or breastfeeding at screening, planning future pregnancies or unwilling to take measures to avoid pregnancy for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in total body weight (in Kg) | 28 weeks
  Between-group differences in percent change from baseline to week 28 in total body weight

SECONDARY OUTCOMES:
Proportion of subjects not achieving 5% weight loss from baseline to week 16 | 16 weeks
  Between-group differences in number of subjects who do not achieve a 5% weight loss (in Kg) from baseline to week 16
Changes in numbers and function of immune cell subsets | 40 weeks
  Between-group differences in percent change from baseline in numbers and functions of immune cells subsets (NK cells, MAIT cells, T-cells and Monocytes) as assessed through flow cytometry in a single assay
Changes in quantified viral reservoir in peripheral blood mononuclear cells (PBMCs) | 40 weeks
  Between-group differences in percent change from baseline in HIV pro-viral DNA and cell-associated RNA (CA-RNA), measured in PBMCs (copies/mL)
Changes in gut microbiome composition in stool samples | 40 weeks
  Between-group differences in percent change from baseline in gut microbiome composition (% prevalence of different microbial species) as assessed through molecular techniques in stool samples
Changes in parameters of glucose metabolism in blood samples | 40 weeks
  Between-group differences in percent change from baseline in blood glucose levels (in mmol/L), HbA1c (in mmol/mol) and insulin levels (in pmol/L)
Changes in parameters of lipid metabolism | 40 weeks
  Between-group differences in percent change from baseline in lipid profile: total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides (all in mmol/L)
Proportion of subjects reporting any adverse event | 40 weeks
  Between-group differences in the number of subjects reporting any type of adverse event, including serious adverse events and suspected unexpected serious adverse reactions
Changes in bone mineral density (BMD) and total body composition | 40 weeks
  Between-group differences in percent change from baseline in lumbar spine and hip BMD and total body composition (% fat mass and lean mass) as assessed through DXA scan
Changes in liver stiffness | 40 weeks
  Between-group differences in percent change from baseline in liver stiffness (measured in kPa) as assessed thourgh liver elastography

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Sullivan L, Savinelli S, O'Hare S, Holden S, McHugh C, Mallon P, Doran P. An enhanced participant information leaflet and multimedia intervention to improve the quality of informed consent to a randomised clinical trial enrolling people living with HIV and obesity: a protocol for a Study Within A Trial (SWAT). Trials. 2022 Jan 17;23(1):50. doi: 10.1186/s13063-021-05979-y. PMID 35039057